CLINICAL TRIAL: NCT02400697
Title: Placental Transfusion in Preterm Infants Born at Less Than 34 Weeks of Gestation … Role of "Delayed" Cord Clamping and Umbilical Cord Milking
Brief Title: Placental Transfusion Project for Preterm Infants
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, William A. Engle, Professor of Pediatrics, Indiana University
Other Study IDs: 1404705195
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Intraventricular Hemorrhage; Sepsis; Necrotizing Enterocolitis
MeSH Terms: conditions — Sepsis; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- <30 wks gestation or 1500 grams: Preterm infants born at participating hospitals
  Interventions: Other: <30 wks gestation or 1500 grams
- 30 wks to <34 wks gestation: Preterm infants born at participating hospitals
  Interventions: Other: <30 wks gestation or 1500 grams

INTERVENTIONS:
Other: <30 wks gestation or 1500 grams — Outcomes of preterm infants recorded

SUMMARY:
The American College of Obstetrics and Gynecology, American Academy of Pediatrics and the World Health Organization have recently published recommendations related to placental transfusions in preterm infants. This project will review outcomes of preterm infants following a quality improvement implementation process in several delivery centers in Indiana. Centers involved in this project are also part of the Indiana Vermont Oxford Network (IRB#1003-84). Data is recorded for that network and the investigators site will be reviewing that data every 3 months from infants who have completed the Vermont Oxford Network collection. This project will specifically look at the incidence of intraventricular hemorrhage, necrotizing entercolitis, periventricular leukomalacia, sepsis and death following the implementation of the ACOG recommendations.

DETAILED DESCRIPTION:
Centers involved in this project are also part of the Indiana Vermont Oxford Network. Data is recorded for that network and the investigators site will be reviewing that data every 3 months from infants who have completed the Vermont Oxford Network collection. This project will specifically look at the incidence of intraventricular hemorrhage, necrotizing entercolitis, periventricular leukomalacia, sepsis and death following the implementation of the ACOG recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born at participating hospital who are less than 30 weeks gestation or less than 1500 grams and/or preterm infants 30 weeks to less than 34 weeks gestation

Exclusion Criteria:

* None

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants less than 30 weeks gestation or less than 1500 grams and/or preterm infants 30 weeks to less than 34 weeks gestation.
Sampling Method: Non-Probability Sample
Enrollment: 2856 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Decrease in common complications of preterm birth | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: William Engle, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States